CLINICAL TRIAL: NCT06822621
Title: Functional Cereal Products and Contribution to the Regulation of Metabolism and Obesity-induced Chronic Low-grade Inflammation-MetaflammationBread
Brief Title: Functional Cereal Products and Contribution to the Regulation of Metabolism and Obesity-induced Chronic Low-grade Inflammation.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Harokopio University (Other)
Collaborators: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Amalia Yanni, Senior Researcher, Harokopio University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 106/2023_16.11.23
Record Dates: First submitted 2025-01-31; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Hypercholesterolemia; Overweight/Obesity
Keywords: hypercholesterolemia; bread; beta-glucans; overweight/obesity; gut microbiota
MeSH Terms: conditions — Hypercholesterolemia; Overweight; Obesity | interventions — Methods

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Dietary intervention with common white wheat bread in mildly hypercholesterolemic subjects with overweight/obesity.
  Interventions: Other: Control
- Intervention group (Active Comparator): Dietary intervention with white wheat bread enriched with oat beta-glucans in mildly hypercholesterolemic subjects with overweight/obesity.
  Interventions: Other: Intervention

INTERVENTIONS:
Other: Control — Dietary intervention with common white wheat bread in mildly hypecholesterolemic subjects following a hypocaloric diet.
  Arms: Control group
Other: Intervention — Dietary intervention with white wheat bread enriched with oat beta-glucans in mildly hypecholesterolemic subjects following a hypocaloric diet.
  Arms: Intervention group

SUMMARY:
The goal of this clinical trial is to find out the possible beneficial effects of a white wheat bread enriched with oat beta-glucans on mildly hypercholesterolemic subjects with overweight/obesity.

The main questions it aims to answer are:

Does the enriched bread lower total and LDL-cholesterol levels as well as the levels of inflammatory factors of the participants? Does the enriched bread positively change the composition of gut microbiota? Researchers will compare the enriched bread to a common white wheat bread to see if the enriched bread provides additional effect beyond a hypocaloric dietary plan that the participants of both groups are going to follow.

Participants will:

Take the enriched or the common bread every day for 8 weeks. Visit the clinic once every 2 weeks for checkups and tests.

DETAILED DESCRIPTION:
The effect of consuming the new bread product, a white wheat bread enriched with oat beta-glucans, on metabolic and inflammatory markers after an 8-week dietary intervention in volunteers with overweight/obesity will be studied. The volunteers will be randomly divided into two groups: group 1 (control) which will receive the conventional product i.e., white wheat bread and group 2 (intervention) which will receive the beta-glucans enriched bread. Both products will be consumed in isocaloric amounts and volunteers in both groups will follow a hypocaloric diet.

The following procedures/determinations will take place at the beginning and end of the intervention:

1. Anthropometric characteristics: weight, height, body mass index (BMI), waist circumference, hip circumference, body composition.
2. Classical biochemical parameters: glycemic control, lipid profile, liver enzymes, urea, creatinine, uric acid.
3. Inflammation status.
4. Estimation of daily energy intake by completing a food consumption frequency questionnaire.
5. Assessment of physical activity.

At the beginning and at the end of the nutritional intervention, stool collection will take place. The samples will be subjected to microbiological and molecular analysis (Next Generation Sequencing, NGS) to determine the microbial populations and the intestinal microbiome.

ELIGIBILITY:
Inclusion Criteria:

* no underlying diseases
* with LDL-cholesterol levels between 115-150 mg/dL
* with 25<BMI<32 kg/m2
* with stable body weight in the last 3 months before the intervention
* with normal diet and exercise habits

Exclusion Criteria:

* not suffer from diabetes mellitus, cardiovascular disease, chronic renal failure
* not receive hypolipidemic treatment
* not receive nutritional supplements that may affect blood lipid levels (eg omega-3 supplements, plant sterols/stanols) or the intestinal microbial flora (probiotics/prebiotics/antibiotics).
* not be pregnant or lactating
* not have food allergies
* not have habits that prevent their compliance with the research protocol

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-02 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Change of serum total- and LDL-cholesterol concentrations of study participants as determined by biochemical analysis | From enrollment to the end of treatment at 8 weeks
  Positive effect of consumption of the bread enriched with beta-gucans in the reduction of total- and LDL-cholesterol concentrations

SECONDARY OUTCOMES:
Change in the composition of gut microbiota as determined by NGS analysis of fecal samples | From enrollment to the end of treatment at 8 weeks.
  Positive effect of consumption of the bread enriched with beta-gucans on the composition of gut microbiota of the study participants

CONTACTS AND LOCATIONS:
Overall Officials: Amalia E Yanni, Senior Researcher, Principal Investigator — Harokopio University; Alexandros Kokkinos, Professor, Study Chair — National and Kapodistrian University of Athens, School of Medicine
Locations (1):
- National and Kapodistrian University of Athens, School of Medicine, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No